CLINICAL TRIAL: NCT03108599
Title: Engineering and Behavioral Controls for Truck Drivers' Sleep, Safety, and Health
Brief Title: Tech4Rest Trial With Team Truck Drivers
Acronym: Tech4Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency); Washington State, Department of Labor and Industries (Unknown); University of Washington (Other)
Responsible Party: Principal Investigator, Ryan Olson, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15440
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Sleep; Sleep Disturbance; Sleep Disorder, Shift Work; Health Knowledge, Attitudes, Practice; Health Behavior; Fatigue; Vibration; Exposure
Keywords: Health Promotion; Injury Prevention; Safety; Wellbeing; Physical Activity; Sleep; Whole Body Vibration; Self-Monitoring
MeSH Terms: conditions — Parasomnias; Sleep Disorders, Circadian Rhythm; Behavior; Health Behavior; Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: In the randomized controlled trial, participants will be randomly assigned to either the control or intervention groups. Following a baseline period, intervention participants will receive the enhanced cab portion of the intervention on its own. Then, for the following intervention phase, intervention participants will participate in the behavioral sleep program in addition to continuing the enhanced cab intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All participants in the intervention arm will receive two interventions: an enhanced cab intervention alone, and then the enhanced cab conditions combined with a behavioral sleep intervention.
  Interventions: Other: Enhanced Cab; Behavioral: Fit4Sleep
- Control (No Intervention): Usual practices with regards to cab conditions and access to workplace programs for preventing sleep and fatigue problems.

INTERVENTIONS:
Other: Enhanced Cab — The enhanced cab intervention includes the introduction of an active suspension seat and a therapeutic mattress system. After a baseline phase, the intervention arm will receive the enhanced cab intervention alone, and then the enhanced cab plus a behavioral sleep program.
  Arms: Intervention
Behavioral: Fit4Sleep — The behavioral sleep program includes a friendly dyad-based physical activity competition; self-monitoring and logging of physical activity, sleep hygiene behaviors, and sleep; and individual coaching. The behavioral sleep program includes an optional body weight management component. The intervention arm will receive the behavioral sleep program in combination with the enhanced cab intervention.
  Other Names: Behavioral Sleep Program
  Arms: Intervention

SUMMARY:
The current project is a safety and health intervention focused on sleep and fatigue among truck driver teams (pairs), where one driver sleeps in a moving vehicle while the other partner drives. This study is conducted within the Oregon Healthy Workforce Center (OHWC), a NIOSH Center of Excellence in Total Worker Health. We will evaluate engineering and behavioral interventions to improve sleep, reduce fatigue, and impact Total Worker Health. An enhanced cab intervention will alter whole body vibrations during driving and sleep periods, and includes a therapeutic mattress system and an active suspension seat. The enhanced cab will be evaluated alone and in combination with a behavioral sleep intervention adapted from our effective SHIFT (Safety &Health Involvement For Truckers) program. The interventions prioritize hazard reduction according to the hierarchy of controls, and will be evaluated with a randomized controlled design.

DETAILED DESCRIPTION:
Total Worker Health® (TWH) is defined as policies, programs, and practices that integrate protection from work-related safety and health hazards with promotion of injury and illness prevention efforts to advance worker well-being. Sleep deficiency is a cross-cutting factor for TWH that not only impacts workplace safety, but also generates excess risk for obesity, chronic disease, and early mortality. Long-haul truck drivers average less sleep per night on the road than they do when sleeping at home due to long, irregular work hours and unfavorable sleeping conditions in truck sleeper berths (e.g., low quality mattresses, vibrations, noise, temperature). Sleep deficiency in trucking is a likely contributor to the 69% prevalence of obesity among US drivers, which increases the risk of obstructive sleep apnea and deadly crashes. Despite the severity of these interacting problems, research on engineering controls in commercial truck cabs to improve sleep and reduce fatigue is limited. Behavioral interventions to improve sleep among truck drivers are also limited. We must address these gaps and evaluate the economic cost-utility of interventions to stimulate industry investment in factors that substantially improve drivers' TWH.

The primary goal of this proposal is to evaluate the effects of an enhanced cab intervention on long-haul truck drivers' sleep and TWH with a randomized controlled design. A secondary goal is to evaluate the additive effects of a behavioral sleep intervention. We focus on truck driver teams (pairs), where one driver sleeps in a moving vehicle while the other partner drives, who experience twice as many awakenings as solo drivers. Our enhanced cab intervention will alter whole body vibrations during driving and sleep periods, and includes a therapeutic mattress system with anti-vibration characteristics (Thevorest) and an active suspension seat (BoseRide III). The enhanced cab will be evaluated alone and in combination with a behavioral sleep intervention adapted from our effective SHIFT program. Our preliminary studies show that the therapeutic mattress system alters vibrations and is strongly preferred by drivers, the active suspension seat reduces vibration exposure and fatigue, and that SHIFT produces robust health behavior changes. Our primary hypotheses are that relative to a control group, the enhanced cab intervention will improve objective measures of (a) sleep duration and quality, (b) fatigue, and (c) driver performance. We will also measure impacts on musculoskeletal pain, well-being, and health behaviors (diet, physical activity). We also hypothesize that intervention effects will be larger when combined with a behavioral sleep intervention. Our propensity for success is bolstered by our unique prior accomplishments and strong trucking industry support. To accomplish our goals and test our hypotheses we propose a 5-year project to accomplish 3 specific aims:

1. Pilot test intervention and experimental procedures. We will conduct formative research with dispatchers and driving teams and adapt our SHIFT intervention to focus explicitly on improving sleep. We will then pilot data collection and intervention procedures (enhanced cab and behavioral interventions) with team truck drivers. This preliminary work will guide adjustments prior to our randomized controlled trial.
2. Determine the effectiveness of an enhanced cab intervention alone and in combination with a behavioral sleep intervention for improving truck drivers' sleep, fatigue, and performance. Teams will be randomized into intervention and control groups. Intervention teams will complete 3 phases: baseline, enhanced cab intervention, and enhanced cab intervention + behavioral sleep intervention. Control teams will be measured at the same time points. Primary outcomes will include sleep duration and quality (actigraphy), fatigue (psychomotor vigilance task), and driver performance (fuel efficiency and hard braking events). Secondary outcomes will include musculoskeletal symptoms, well-being, diet, and exercise.
3. Conduct cost-utility analyses for interventions. We will gather historical data from trucking companies and model the cost-utility of intervention components. Model variables will include intervention costs and estimated returns or savings based on intervention effects, such as improvements in driver performance (e.g., fuel efficiency), reduced lost workdays, and reduced probability of fatigue-related crashes.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a team truck driver with a driving partner who is also willing to participate.
* Employed at a company that supports the project requirements

Exclusion Criteria:

* Non-treatment compliant for diagnosed Obstructive Sleep Apnea
* Driving teammate is unwilling, unable, or ineligible to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-reported sleep duration in hours at 2 months | Baseline and 2 months (post-enhanced cab)
  Pittsburgh Sleep Quality Index sleep duration question (more hours is better sleep duration)
Change from baseline in self-reported sleep duration in hours at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Pittsburgh Sleep Quality Index sleep duration question (more hours is better sleep duration)
Change from baseline in self-reported sleep quality at 2 months | Baseline and 2 months (post-enhanced cab)
  Pittsburgh Sleep Quality Index sleep quality question (0-3, higher is better sleep quality)
Change from baseline in self-reported sleep quality at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Pittsburgh Sleep Quality Index sleep quality question (0-3, higher is better sleep quality)
Change from baseline in sleep disturbance at 2 months | Baseline and 2 months (post-enhanced cab)
  Sleep Disturbance Scale, Patient-Reported Outcomes Measurement Information System (8-40, higher is worse [greater sleep disturbance])
Change from baseline in sleep-related impairment at 2 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Sleep Disturbance Scale, Patient-Reported Outcomes Measurement Information System (8-40, higher is worse [greater sleep disturbance])
Change from baseline in sleep-related impairment at 2 months | Baseline and 2 months (post-enhanced cab)
  Sleep-Related Impairment Scale, Patient-Reported Outcomes Measurement Information System (8-40, higher is worse [greater sleep-related impairment])
Change from baseline in sleep-related impairment at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Sleep-Related Impairment Scale, Patient-Reported Outcomes Measurement Information System (8-40, higher is worse [greater sleep-related impairment])
Change from baseline in self-reported fatigue at 2 months | Baseline and 2 months (post-enhanced cab)
  Swedish Occupational Fatigue Inventory (0-48, higher is worse [more fatigue])
Change from baseline in self-reported fatigue at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program
  Swedish Occupational Fatigue Inventory (0-48, higher is worse [more fatigue])
Change from baseline in actigraphic measures of sleep duration in hours at 2 months | One week samples at Baseline and 2 months (post-enhanced cab)
  Direct measurement via Actigraph GT3x+ BT (more hours is better sleep duration)
Change from baseline in actigraphic measures of sleep duration in hours at 3-4 months | One week samples at Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Actigraph GT3x+ BT (more hours is better sleep duration)
Change from baseline in actigraphic measures of sleep efficiency percentage at 2 months | One week samples at Baseline and 2 months (post-enhanced cab)
  Direct measurement via Actigraph GT3x+ BT (higher percentage is better sleep efficiency)
Change from baseline in actigraphic measures of sleep efficiency percentage at 3-4 months | One week samples at Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Actigraph GT3x+ BT (higher percentage is better sleep efficiency)

SECONDARY OUTCOMES:
Change from baseline in sleep hygiene practices at 2 months | Baseline and 2 months (post-enhanced cab)
  Sleep Hygiene Index (0-48, higher is worse sleep hygiene)
Change from baseline in sleep hygiene practices at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Sleep Hygiene Index (0-48, higher is worse sleep hygiene)
Change from baseline in self-reported days per week with moderate intensity physical activity at 2 months | Baseline and 2 months (post-enhanced cab)
  International Physical Activity Scale-Short Form moderate intensity physical activity question (0-7 days, more days is better moderate physical activity levels)
Change from baseline in self-reported moderate intensity physical activity at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  International Physical Activity Scale-Short Form moderate intensity physical activity question (0-7 days, more days is better moderate physical activity levels)
Change from baseline in self-reported vigorous intensity physical activity at 2 months | Baseline and 2 months (post-enhanced cab)
  International Physical Activity Scale-Short Form vigorous physical activity question (0-7 days, more days is better vigorous intensity physical activity levels)
Change from baseline in self-reported vigorous intensity physical activity at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  International Physical Activity Scale-Short Form vigorous physical activity question (0-7 days, more days is better vigorous intensity physical activity levels)
Change from baseline in actigraphy measures of minutes per week in physical activity bouts at 2 months | One week samples at Baseline and 2 months (post-enhanced cab)
  Direct measurement via Actigraph GT3x+ BT (more minutes is better)
Change from baseline in actigraphy measures of minutes per week in physical activity bouts at 3-4 months | One week samples at Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Actigraph GT3x+ BT (more minutes is better)
Change from baseline in actigraphy measures of 10-minute physical activity bouts at 2 months | One week samples at Baseline and 2 months (post-enhanced cab)
  Direct measurement via Actigraph GT3x+ BT (more bouts is better)
Change from baseline in actigraphy measures of 10-minute physical activity bouts at 3-4 months | One week samples at Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Actigraph GT3x+ BT (more bouts is better)
Change from baseline in well-being (physical health) at 2 months | Baseline and 2 months (post-enhanced cab)
  Physical Health Subscale of the Patient-Reported Outcomes Measurement Information System Global Health Scale (4-20, higher is better physical health)
Change from baseline in well-being (physical health) at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Physical Health Subscale of the Patient-Reported Outcomes Measurement Information System Global Health Scale (4-20, higher is better physical health)
Change from baseline in well-being (mental health) at 2 months | Baseline and 2 months (post-enhanced cab)
  Mental Health Subscale of the Patient-Reported Outcomes Measurement Information System Global Health Scale (4-20, higher is better mental health)
Change from baseline in well-being (mental health) at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Mental Health Subscale of the Patient-Reported Outcomes Measurement Information System Global Health Scale (4-20, higher is better mental health)

OTHER OUTCOMES:
Change from baseline in body weight at 2 months | Baseline and 2 months (post-enhanced cab)
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer (higher weight is worse)
Change from baseline in body weight at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer (higher weight is worse)
Change from baseline in body mass index at 2 months | Baseline and 2 months (post-enhanced cab)
  Direct measurement via stadiometer and Tanita TBF-310GS Bioelectric Impedance Analyzer (higher body mass index is worse)
Change from baseline in body mass index at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via stadiometer and Tanita TBF-310GS Bioelectric Impedance Analyzer (higher body mass index is worse)
Change from baseline in percent body fat at 2 months | Baseline and 2 months (post-enhanced cab)
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer (higher percent body fat is worse)
Change from baseline in percent body fat at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Tanita TBF-310GS Bioelectric Impedance Analyzer (higher percent body fat is worse)
Change from baseline in systolic blood pressure at 2 months | Baseline and 2 months (post-enhanced cab)
  Direct measurement via Omron HEM-907 automatic blood pressure monitor (higher systolic blood pressure is worse)
Change from baseline in systolic blood pressure at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Omron HEM-907 automatic blood pressure monitor (higher systolic blood pressure is worse)
Change from baseline in diastolic blood pressure at 2 months | Baseline and 2 months (post-enhanced cab)
  Direct measurement via Omron HEM-907 automatic blood pressure monitor (higher diastolic blood pressure is worse)
Change from baseline in diastolic blood pressure at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Direct measurement via Omron HEM-907 automatic blood pressure monitor (higher diastolic blood pressure is worse)
Change from baseline in fruit and vegetable servings per day at 2 months | Baseline and 2 months (post-enhanced cabs)
  Single-item on number of fruit and vegetable servings developed by investigators (0-5+, more servings is better)
Change from baseline in fruit and vegetable servings per day at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Single-item on number of fruit and vegetable servings developed by investigators (0-5+, more servings is better)
Change from baseline in frequency of meals brought from home at 2 months | Baseline and 2 months (post-enhanced cab)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of meals brought from home at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of consumption of sugary snacks at 2 months | Baseline and 2 months (post-enhanced cab)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of consumption of sugary snacks at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of sugary drink consumption at 2 months | Baseline and 2 months (post-enhanced cab)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of sugary drink consumption at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of fast food consumption at 2 months | Baseline and 2 months (post-enhanced cab)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in frequency of fast food consumption at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  single item from prior research by other investigators (0 [Never] to 9 [5 or more times per day], higher is better)
Change from baseline in pain interference with home and work activities at 2 months | Baseline and 2 months (post-enhanced cab)
  Adapted Nordic-style questionnaire for musculoskeletal symptoms (5-25, higher is worse [greater pain interference])
Change from baseline in pain interference with home and work activities at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Adapted Nordic-style questionnaire for musculoskeletal symptoms (5-25, higher is worse [greater pain interference])
Change from baseline in pain intensity at 2 months | Baseline and 2 months (post-enhanced cab)
  Adapted Nordic-style questionnaire for musculoskeletal symptoms (0-50, higher is worse pain)
Change from baseline in pain intensity at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Adapted Nordic-style questionnaire for musculoskeletal symptoms (0-50, higher is worse pain)
Change from baseline in driving vehicle collisions without damage at 2 months | Baseline and 2 months (post-enhanced cab)
  Self-reported vehicle collisions without damage using item created by investigators (0-5+, more is worse)
Change from baseline in driving vehicle collisions without damage at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Self-reported vehicle collisions without damage using item created by investigators (0-5+, more is worse)
Change from baseline in driving vehicle collisions with damage at 2 months | Baseline and 2 months (post-enhanced cab)
  Self-reported vehicle collisions with damage using two items created by investigators (0-5+, more is worse)
Change from baseline in driving vehicle collisions with damage at 2 and 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Self-reported vehicle collisions with damage using two items created by investigators (0-5+, more is worse)
Change from baseline in minor injuries at work at 2 months | Baseline and 2 months (post-enhanced cab)
  Self-reported worker injuries without lost work time using item created by investigators (0-5+, more is worse)
Change from baseline in minor injuries at work at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Self-reported worker injuries without lost work time using item created by investigators (0-5+, more is worse)
Change from baseline in major injuries at work at 2 months | Baseline and 2 months (post-enhanced cab)
  Self-reported worker injuries resulting in lost work time using item created by investigators (0-5+, more is worse)
Change from baseline in major injuries at work at 3-4 months | Baseline and 3-4 months (post-enhanced cab + behavioral sleep program)
  Self-reported worker injuries resulting in lost work time using item created by investigators (0-5+, more is worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared with researchers outside of the primary research team. De-identified data will be shared only after receiving IRB approval.

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Ahsberg E. Dimensions of fatigue in different working populations. Scand J Psychol. 2000 Sep;41(3):231-41. doi: 10.1111/1467-9450.00192. PMID 11041305
- [Background] Mastin DF, Bryson J, Corwyn R. Assessment of sleep hygiene using the Sleep Hygiene Index. J Behav Med. 2006 Jun;29(3):223-7. doi: 10.1007/s10865-006-9047-6. Epub 2006 Mar 24. PMID 16557353
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Buxton OM, Quintiliani LM, Yang MH, Ebbeling CB, Stoddard AM, Pereira LK, Sorensen G. Association of sleep adequacy with more healthful food choices and positive workplace experiences among motor freight workers. Am J Public Health. 2009 Nov;99 Suppl 3(Suppl 3):S636-43. doi: 10.2105/AJPH.2008.158501. PMID 19890169
- [Background] Dennerlein JT, Hopcia K, Sembajwe G, Kenwood C, Stoddard AM, Tveito TH, Hashimoto DM, Sorensen G. Ergonomic practices within patient care units are associated with musculoskeletal pain and limitations. Am J Ind Med. 2012 Feb;55(2):107-16. doi: 10.1002/ajim.21036. Epub 2011 Nov 23. PMID 22113975
- [Background] Hedge A, Morimoto S, McCrobie D. Effects of keyboard tray geometry on upper body posture and comfort. Ergonomics. 1999 Oct;42(10):1333-49. doi: 10.1080/001401399184983. PMID 10582503
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Result] Olson R, Johnson PW, Shea SA, Marino M, Springer R, Rice SPM, Rimby J, Donovan C. The Tech4Rest Randomized Controlled Trial: Applying the Hierarchy of Controls to Advance the Sleep, Health, and Well-being of Team Truck Drivers. J Occup Environ Med. 2023 Nov 1;65(11):937-948. doi: 10.1097/JOM.0000000000002941. Epub 2023 Aug 12. PMID 37590443